CLINICAL TRIAL: NCT02925182
Title: Treatment of Recurrent Aphthous Stomatitis With Er,Cr:YSGG Laser Irradiation: A Randomized Controlled Clinical Study
Brief Title: Treatment of Recurrent Aphthous Stomatitis With Er,Cr:YSGG Laser Irradiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Hasan Guney YILMAZ, Assoc Prof Dr, Near East University, Turkey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CE018-2015
Record Dates: First submitted 2016-09-28; First posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Stomatitis, Aphthous
MeSH Terms: conditions — Stomatitis, Aphthous

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- test (Experimental): Recurrent Aphthous Stomatitis were irradiated with Er,Cr:YSGG laser (Waterlase MD, Biolase, Irvine, CA, USA) on hard tissue mode with a mg6 sapphire tip (600 µm diameter, 6 mm length) using non-contact mode at an energy level of 0.25W and a repetition rate of 20 kHz and pulse duration of 140 µs, 0% water and 10% air at 5 J/cm2 energy density. The treatment time was 20 s per surface by scanning the Recurrent Aphthous Stomatitis area.
  Interventions: Device: Er,Cr:YSGG Laser
- Control (Placebo Comparator): In the placebo group, the same Er,Cr:YSGG laser without laser emission was used.
  Interventions: Device: Er,Cr:YSGG Laser

INTERVENTIONS:
Device: Er,Cr:YSGG Laser
  Other Names: Waterlase MD

SUMMARY:
The aim this study was to investigate the efficacy of Er,Cr:YSGG laser irradiation in reducing pain and on healing rate of recurrent aphthous stomatitis 40 patients with RAS were included to the study. For each patient, ulceration were randomly assigned to the test or the control group. In test group RAS irradiated with Er,Cr:YSGG laser using non-contact mode. In the placebo group, the same Er,Cr:YSGG laser without laser emission was used. Pain was evaluated with visual analog scale (VAS). Healing of RAS (HRAS) was graded by a clinician.

ELIGIBILITY:
Inclusion Criteria:

* For inclusion every patient had to have one pairs of minor RAS duration of 3 days or less, in the buccal or labial nonkeratinized oral mucosa.

Exclusion Criteria:

* Patients with a known systemic disease that predisposed them to RAS (e.g., Behçet disease), presence of any major herpetic lesions, traumatic ulcers, ulcers caused due to topical or systemic medications, or undergoing systemic or local treatment for RAS were excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Reduce of Visual Analog Scale (VAS) scores | 10 days
  Patients were asked to record their pain and discomfort level for each stomatit by marking a point on a 10 cm visual analog scale (VAS).

SECONDARY OUTCOMES:
The healing of recurrent aphthous (HRAS) scores | 10 days
  The healing of RAS (HRAS) were evaluated:at the follow-up sessions by the investigator on a four-point scale (range 1-4). Grade 1 represented totally healing, grade 2 moderate healing (more than 50% of RAS was epithelialized and healed), grade 3 slightly healing (less than 50% of RAS was epithelialized and healed) and grade 4 no healing.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Guney YILMAZ, DDS, PhD, Study Director — Near Easat University, Faculty of Dentistry

IPD SHARING:
Plan to Share IPD: No